CLINICAL TRIAL: NCT06972251
Title: Tailored Approaches to Reduce Distress and Improve Self-Management for Veterans With Diabetes (TARDIS) - Photo Elicitation and Intervention
Brief Title: TARDIS - Photo Elicitation and Intervention
Acronym: TARDIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NRI 18-234-1
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type II; Type 2 Diabetes; Diabetes Distress; Self Management; Veteran
Keywords: Diabetes; Type 2 Diabetes; Diabetes distress; Veteran
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aim 3a - TARDIS Photo Elicitation (Other): To further understand Diabetes Distress (DD) by expanding on what we have learned thus far in cognitive and semi-structured interviews with Veterans. Visual-based qualitative methods will help identify and more robustly describe DD in Veterans.
  Interventions: Behavioral: TARDIS Photo Elicitation
- Aim 3b - TARDIS Intervention (Other): Design & pilot test an innovative, tailored self-management information and supportive services intervention for Veterans with type 2 diabetes (T2D), to promote engagement in self-management behaviors.
  Interventions: Behavioral: TARDIS Intervention

INTERVENTIONS:
Behavioral: TARDIS Photo Elicitation — Using visual-based qualitative methods to help identify and more robustly describe DD in Veterans.
  Arms: Aim 3a - TARDIS Photo Elicitation
Behavioral: TARDIS Intervention — Design & pilot test an innovative, tailored self-management information and supportive services intervention for Veterans with type 2 diabetes (T2D), to promote engagement in self-management behaviors.
  Arms: Aim 3b - TARDIS Intervention

SUMMARY:
Veterans with type 2 diabetes (T2D) may become overwhelmed with the self-management behaviors needed to maintain optimal health. Veterans may experience diabetes distress (DD), a concept distinct from depression, due the amount and frequency of these behaviors. Diabetes distress negatively influences the Veteran's engagement in self-management and subsequent glycosylated hemoglobin (HbA1c) levels. Previous interventions aimed at improving T2D self-management and reducing DD do not tailor T2D self-management information to a Veteran's DD, which may be one reason interventions are ineffective at reducing DD.

The purpose of this study is to further understand DD by expanding on what the investigators have learned thus far in cognitive and semi-structured interviews with Veterans (see ClinicalTrials.gov identifier NCT04587336). In Aim 3a, the photo elicitation study, the Veteran would be provided with a camera and instructed to take approximately 20 photos over two weeks. The investigators would conduct two semi-structured interviews with the Veteran to discuss this experience. Visual-based qualitative methods will help us identify and more robustly describe DD in Veterans. In Aim 3b, the investigators will conduct a pilot study of a novel telemedicine intervention.

The TARDIS intervention (Aim 3b) will build off data collected in Aim 3a and provide tailored coaching to Veterans with type 2 diabetes mellitus. The TARDIS intervention includes coaching, self-management information, and referrals to Veterans Health Administration (VHA) supportive services delivered via the telephone. TARDIS will augment current VHA care for patients with diabetes. All Veterans will continue to receive care from their primary clinicians during the study.

DETAILED DESCRIPTION:
Background and Significance: An estimated 20-25% of Veterans are diagnosed with diabetes, an incidence three times higher than the national rate. Treatment and management of poorly self-managed diabetes is costly as medical care costs are 2.3 times higher for individuals with diabetes than for those who do not have the disease. Regular preventative care is essential to prevent comorbidities and maintain optimal health. Individuals with T2D provide 99% of their own care; self-management of T2D is person-specific and ever-present. Consistent and sustained self-management decreases comorbidity development, and positively influences quality of life and psychosocial outcomes. Inconsistent self-management increases the risk of poor health outcomes including microvascular and/or macrovascular problems and psychosocial complications. Yet rates of self-management remain sub-optimal.

T2D self-management is omnipresent, inescapable, and burdensome. A Veteran may become overwhelmed and/or frustrated because of the amount and frequency of T2D self-management behaviors, and these negative feelings may lead to inattention to critical self-management behaviors such as eating healthy or blood glucose checks. Veterans often experience challenges to self-management despite knowing the importance of these behaviors. Self-management challenges include limited access to a healthcare provider, unreliable transportation, limited knowledge of healthy food options, beliefs about T2D medications, or a lack of support. Additionally, diabetes distress (DD) and other psychosocial factors (i.e., depression, post-traumatic stress disorder) negatively influence an individual's engagement in self-management and health outcomes. Due to the inherent complexity of T2D self-management, the investigators propose that tailoring on DD is one way to focus the provision of tailored self-management information and connections to supportive services. Diabetes distress encompasses the cognitive, physical, and affective experience of living with T2D. Diabetes distress occurs when an individual is overwhelmed with T2D, related self-management behaviors, and knowledge that T2D is progressive and incurable. Diabetes distress is subjective and person-specific; and while DD may fluctuate over time, DD may be continually present. Undiagnosed and untreated DD, may be one cause of a Veteran's poor self-management, thus resulting in poor health outcomes.

Diabetes distress is commonly assessed via the Diabetes Distress Scale or the Problem Areas in Diabetes Scale. Research indicates both measures demonstrate the construct of DD is distinct from general anxiety, stress, and depression. Both the Diabetes Distress Scale and Problem Areas in Diabetes scales assess DD in several domains, and each DD domain addresses a separate aspect of the burden of T2D. The Diabetes Distress Scale measures DD in four domains (i.e., regimen, emotional, interpersonal, healthcare provider), and the Problem Areas in Diabetes Scale assesses DD using similar domains (i.e., emotional, diabetes management, treatment, and social support burden). The Diabetes Distress Scale and Problem Areas in Diabetes Scale have demonstrated content validity in measuring an individual's perception of the resources available, or not available, for self-management. Diabetes distress is associated with more T2D complications, increased stress, being prescribed insulin by a healthcare provider, poor diet and exercise, inadequate support environments, and is more prevalent among women. Diabetes distress levels correlate with self-management behaviors such as monitoring one's diet, engaging with providers, and monitoring one's blood glucose. High to moderate levels of DD are related to poorer glucose regulation, higher HbA1c, lower medication adherence, and poorer quality of life. Individuals with DD report diabetes-related physical burden, health care system distress, and distress with comorbid conditions. In this study, the investigators will further examine the Veteran's experience of DD.

The TARDIS grant and the prior work done for TARDIS was based upon the original Diabetes Distress Scale (DDS) and the four domains within that scale. Those domains include: regimen, provider, interpersonal, and emotional. In 2022, the authors of the Diabetes Distress Scale published an updated version of the DDS called the Type 2 Diabetes Distress Assessment System (T2D-DDAS). The T2D-DDAS contains core and source items that contribute to DD. The T2D-DDAS sources include: hypoglycemia, long-term health, health care provider, interpersonal issues, shame/stigma, healthcare access, and management demands. The sources or facets of DD the investigators identified in the TARDIS foundational work are reflected in the T2D-DDAS. Of note, the investigators identified several additional facets of DD in our work such as pain, military experience, living with comorbidities, and being a caregiver. The scoring for low, moderate, and high DD in the DDS and the T2D-DDAS is the same. For the TARDIS intervention, the investigators will be focusing on the domains of DD as measured by the DDS and not the sources of DD as measured by the T2D-DDAS. The DDS is in the Cerner electronic health record (EHR) and is being used in the VA and the foundational TARDIS work uses the DDS.

Aim 3a: Visual Based Qualitative Methods Visual-based qualitative methods will help us identify and more robustly describe DD in Veterans and will expand on what the investigators have learned thus far in cognitive and semi-structured interviews. Veterans will have the autonomy to select photos that impact, either positively or negatively, their DD and diabetes self-management behaviors. Veterans who participate in the project may want to share their experiences because this is their personal story which they want to share to help other people. The Veteran has the autonomy to decide what, and how much, information to share.

Aim 3b: TARDIS Intervention The TARDIS intervention builds upon data collected in Aim 3a. Health coaching is a person-centered approach to identifying health goals, challenges to these goals, and then developing strategies to address these challenges. For the purposes of TARDIS, interactions are 1:1 between a 'coach', or someone who has received training in motivational interviewing, and a Veteran with type 2 diabetes mellitus (T2DM). This personalized approach can help elicit, understand, and address the experience of DD, and its impact on T2DM self-management, in Veterans with T2DM. With personalized, Veteran-centric information and support, a Veteran may be more equipped to implement self-management to overcome his/her personal modifiable challenges to engaging in T2DM self-management.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes (ICD-10 codes: E11.9, E11.8)
* Documentation of HbA1c drawn within the past 180 days
* Able to speak and read English
* Be able to provide informed consent to participate in the study
* Own a mobile phone with advanced computing capabilities (otherwise known as a smartphone) or mobile device to take photos (Aim 3a only)
* hemoglobin A1C (HbA1C) test value greater than or equal to 8.5 (Aim 3b only)
* Be prescribed insulin (Aim 3b only)

Exclusion Criteria:

* New diagnosis of T2D within the last 60 days
* Hospitalization for mental illness within the past 30 days
* Receiving active chemotherapy and/or radiation treatment
* Diagnosis for metastatic cancer
* Recent hospitalization within the past 60 days that would influence their diabetes medication regimen (e.g., myocardial infarction, cerebrovascular accident, coronary artery bypass grafting, etc.)
* Currently receiving kidney dialysis
* Limited hearing or speech difficulties that influence the Veteran's ability to complete the survey and intervention
* Dementia, delirium, or other cognition issues that influence the Veteran's ability to provide consent and complete the survey
* Not currently prescribed insulin (Aim 3b only)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allison Lewinski, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Veterans Health Administration. VA Research on Diabetes. Atlanta, GA.: U.S. Department of Veterans Affairs, Veterans Health Administration, Office of Research and Development; 2016: https://www.research.va.gov/pubs/docs/va_factsheets/Diabetes.pdf.
- [Background] American Diabetes Association. Economic Costs of Diabetes in the U.S. in 2017. Diabetes Care. 2018 May;41(5):917-928. doi: 10.2337/dci18-0007. Epub 2018 Mar 22. PMID 29567642
- [Background] Funnell MM, Anderson RM. Working toward the next generation of diabetes self-management education. Am J Prev Med. 2002 May;22(4 Suppl):3-5. doi: 10.1016/s0749-3797(02)00431-2. No abstract available. PMID 11985929
- [Background] Norris SL, Lau J, Smith SJ, Schmid CH, Engelgau MM. Self-management education for adults with type 2 diabetes: a meta-analysis of the effect on glycemic control. Diabetes Care. 2002 Jul;25(7):1159-71. doi: 10.2337/diacare.25.7.1159. PMID 12087014
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Ahola AJ, Groop PH. Barriers to self-management of diabetes. Diabet Med. 2013 Apr;30(4):413-20. doi: 10.1111/dme.12105. PMID 23278342
- [Background] Laranjo L, Neves AL, Costa A, Ribeiro RT, Couto L, Sa AB. Facilitators, barriers and expectations in the self-management of type 2 diabetes--a qualitative study from Portugal. Eur J Gen Pract. 2015 Jun;21(2):103-10. doi: 10.3109/13814788.2014.1000855. Epub 2015 Feb 20. PMID 25698085
- [Background] Gariepy G, Smith KJ, Schmitz N. Diabetes distress and neighborhood characteristics in people with type 2 diabetes. J Psychosom Res. 2013 Aug;75(2):147-52. doi: 10.1016/j.jpsychores.2013.05.009. Epub 2013 Jul 3. PMID 23915771
- [Background] Tanenbaum ML, Kane NS, Kenowitz J, Gonzalez JS. Diabetes distress from the patient's perspective: Qualitative themes and treatment regimen differences among adults with type 2 diabetes. J Diabetes Complications. 2016 Aug;30(6):1060-8. doi: 10.1016/j.jdiacomp.2016.04.023. Epub 2016 May 4. PMID 27217023
- [Background] Fisher L, Hessler D, Glasgow RE, Arean PA, Masharani U, Naranjo D, Strycker LA. REDEEM: a pragmatic trial to reduce diabetes distress. Diabetes Care. 2013 Sep;36(9):2551-8. doi: 10.2337/dc12-2493. Epub 2013 Jun 4. PMID 23735726
- [Background] Anderson RJ, Freedland KE, Clouse RE, Lustman PJ. The prevalence of comorbid depression in adults with diabetes: a meta-analysis. Diabetes Care. 2001 Jun;24(6):1069-78. doi: 10.2337/diacare.24.6.1069. PMID 11375373
- [Background] Aronson BD, Palombi LC, Walls ML. Rates and consequences of posttraumatic distress among American Indian adults with type 2 diabetes. J Behav Med. 2016 Aug;39(4):694-703. doi: 10.1007/s10865-016-9733-y. Epub 2016 Mar 21. PMID 27001254
- [Background] Aikens JE, Zivin K, Trivedi R, Piette JD. Diabetes self-management support using mHealth and enhanced informal caregiving. J Diabetes Complications. 2014 Mar-Apr;28(2):171-6. doi: 10.1016/j.jdiacomp.2013.11.008. Epub 2013 Nov 27. PMID 24374137
- [Background] Fisher L, Hessler DM, Polonsky WH, Mullan J. When is diabetes distress clinically meaningful?: establishing cut points for the Diabetes Distress Scale. Diabetes Care. 2012 Feb;35(2):259-64. doi: 10.2337/dc11-1572. Epub 2012 Jan 6. PMID 22228744
- [Background] Adriaanse MC, Pouwer F, Dekker JM, Nijpels G, Stehouwer CD, Heine RJ, Snoek FJ. Diabetes-related symptom distress in association with glucose metabolism and comorbidity: the Hoorn Study. Diabetes Care. 2008 Dec;31(12):2268-70. doi: 10.2337/dc08-1074. Epub 2008 Aug 26. PMID 18728236
- [Background] Welch GW, Jacobson AM, Polonsky WH. The Problem Areas in Diabetes Scale. An evaluation of its clinical utility. Diabetes Care. 1997 May;20(5):760-6. doi: 10.2337/diacare.20.5.760. PMID 9135939
- [Background] Schmitt A, Reimer A, Kulzer B, Haak T, Ehrmann D, Hermanns N. How to assess diabetes distress: comparison of the Problem Areas in Diabetes Scale (PAID) and the Diabetes Distress Scale (DDS). Diabet Med. 2016 Jun;33(6):835-43. doi: 10.1111/dme.12887. Epub 2015 Sep 8. PMID 26287511
- [Background] Fisher L, Glasgow RE, Strycker LA. The relationship between diabetes distress and clinical depression with glycemic control among patients with type 2 diabetes. Diabetes Care. 2010 May;33(5):1034-6. doi: 10.2337/dc09-2175. Epub 2010 Feb 11. PMID 20150291
- [Background] Baek RN, Tanenbaum ML, Gonzalez JS. Diabetes burden and diabetes distress: the buffering effect of social support. Ann Behav Med. 2014 Oct;48(2):145-55. doi: 10.1007/s12160-013-9585-4. PMID 24550072
- [Background] Berry E, Lockhart S, Davies M, Lindsay JR, Dempster M. Diabetes distress: understanding the hidden struggles of living with diabetes and exploring intervention strategies. Postgrad Med J. 2015 May;91(1075):278-83. doi: 10.1136/postgradmedj-2014-133017. Epub 2015 Mar 31. PMID 25827438
- [Background] Dennick K, Sturt J, Speight J. What is diabetes distress and how can we measure it? A narrative review and conceptual model. J Diabetes Complications. 2017 May;31(5):898-911. doi: 10.1016/j.jdiacomp.2016.12.018. Epub 2017 Feb 14. PMID 28274681
- [Background] Chesla CA, Chun KM, Kwan CM, Mullan JT, Kwong Y, Hsu L, Huang P, Strycker LA, Shum T, To D, Kao R, Waters CM. Testing the efficacy of culturally adapted coping skills training for Chinese American immigrants with type 2 diabetes using community-based participatory research. Res Nurs Health. 2013 Aug;36(4):359-72. doi: 10.1002/nur.21543. Epub 2013 Apr 19. PMID 23606271
- [Background] Carolan M, Holman J, Ferrari M. Experiences of diabetes self-management: a focus group study among Australians with type 2 diabetes. J Clin Nurs. 2015 Apr;24(7-8):1011-23. doi: 10.1111/jocn.12724. Epub 2014 Nov 3. PMID 25363710
- [Background] Fisher L, Mullan JT, Skaff MM, Glasgow RE, Arean P, Hessler D. Predicting diabetes distress in patients with Type 2 diabetes: a longitudinal study. Diabet Med. 2009 Jun;26(6):622-7. doi: 10.1111/j.1464-5491.2009.02730.x. PMID 19538238
- [Background] Faber-Wildeboer AT, van Os-Medendorp H, Kooy A, Sol BGM. Prevalence and risk factors of depression and diabetes-related emotional distress in patients with type 2 diabetes: A cross-sectional study. Journal of Nursing Education & Practice. 2013;3(6):61-69.
- [Background] Lipscombe C, Smith KJ, Gariepy G, Schmitz N. Gender differences in the association between lifestyle behaviors and diabetes distress in a community sample of adults with type 2 diabetes. J Diabetes. 2016 Mar;8(2):269-78. doi: 10.1111/1753-0407.12298. Epub 2015 May 6. PMID 25850582
- [Background] Perrin NE, Davies MJ, Robertson N, Snoek FJ, Khunti K. The prevalence of diabetes-specific emotional distress in people with Type 2 diabetes: a systematic review and meta-analysis. Diabet Med. 2017 Nov;34(11):1508-1520. doi: 10.1111/dme.13448. Epub 2017 Aug 31. PMID 28799294
- [Background] Sturt, J., Dennick, K., Hessler, D., Hunter, B. M., Oliver, J., & Fisher, L. (2015). Effective interventions for reducing diabetes distress: systematic review and meta-analysis. International Diabetes Nursing, 12(2), 40-55. https://doi.org/10.1179/2057332415Y.0000000004
- [Background] Dennick, K., Sturt, J., Hessler, D., Purssell, E., Hunter, B., Oliver, J., & Fisher, L. (2015). High rates of elevated diabetes distress in research populations: A systematic review and meta-analysis. International Diabetes Nursing, 12(3), 93-107. https://doi.org/10.1080/20573316.2016.1202497
- [Background] Chew BH, Vos RC, Pouwer F, Rutten GEHM. The associations between diabetes distress and self-efficacy, medication adherence, self-care activities and disease control depend on the way diabetes distress is measured: Comparing the DDS-17, DDS-2 and the PAID-5. Diabetes Res Clin Pract. 2018 Aug;142:74-84. doi: 10.1016/j.diabres.2018.05.021. Epub 2018 May 24. PMID 29802952
- [Background] Carper MM, Traeger L, Gonzalez JS, Wexler DJ, Psaros C, Safren SA. The differential associations of depression and diabetes distress with quality of life domains in type 2 diabetes. J Behav Med. 2014 Jun;37(3):501-10. doi: 10.1007/s10865-013-9505-x. Epub 2013 Mar 21. PMID 23515932
- [Background] Polonsky WH, Fisher L, Earles J, Dudl RJ, Lees J, Mullan J, Jackson RA. Assessing psychosocial distress in diabetes: development of the diabetes distress scale. Diabetes Care. 2005 Mar;28(3):626-31. doi: 10.2337/diacare.28.3.626. PMID 15735199
- [Background] Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. Med Care. 2003 Nov;41(11):1284-92. doi: 10.1097/01.MLR.0000093487.78664.3C. PMID 14583691
- [Background] Prins A, Bovin MJ, Smolenski DJ, Marx BP, Kimerling R, Jenkins-Guarnieri MA, Kaloupek DG, Schnurr PP, Kaiser AP, Leyva YE, Tiet QQ. The Primary Care PTSD Screen for DSM-5 (PC-PTSD-5): Development and Evaluation Within a Veteran Primary Care Sample. J Gen Intern Med. 2016 Oct;31(10):1206-11. doi: 10.1007/s11606-016-3703-5. Epub 2016 May 11. PMID 27170304
- [Background] Billioux, A., K. Verlander, S. Anthony, and D. Alley. 2017. Standardized Screening for Health-Related Social Needs in Clinical Settings: The Accountable Health Communities Screening Tool. NAM Perspectives. Discussion Paper, National Academy of Medicine, Washington, DC. https://doi.org/10.31478/201705b
- [Background] Anderson RM, Fitzgerald JT, Gruppen LD, Funnell MM, Oh MS. The Diabetes Empowerment Scale-Short Form (DES-SF). Diabetes Care. 2003 May;26(5):1641-2. doi: 10.2337/diacare.26.5.1641-a. No abstract available. PMID 12716841
- [Background] Kerfoot BP, Gagnon DR, McMahon GT, Orlander JD, Kurgansky KE, Conlin PR. A Team-Based Online Game Improves Blood Glucose Control in Veterans With Type 2 Diabetes: A Randomized Controlled Trial. Diabetes Care. 2017 Sep;40(9):1218-1225. doi: 10.2337/dc17-0310. Epub 2017 Aug 8. PMID 28790131
- [Background] Toobert DJ, Hampson SE, Glasgow RE. The summary of diabetes self-care activities measure: results from 7 studies and a revised scale. Diabetes Care. 2000 Jul;23(7):943-50. doi: 10.2337/diacare.23.7.943. PMID 10895844
- [Background] Weinger K, Butler HA, Welch GW, La Greca AM. Measuring diabetes self-care: a psychometric analysis of the Self-Care Inventory-Revised with adults. Diabetes Care. 2005 Jun;28(6):1346-52. doi: 10.2337/diacare.28.6.1346. PMID 15920050
- [Background] Molina Y, Choi SW, Cella D, Rao D. The stigma scale for chronic illnesses 8-item version (SSCI-8): development, validation and use across neurological conditions. Int J Behav Med. 2013 Sep;20(3):450-60. doi: 10.1007/s12529-012-9243-4. PMID 22639392
- [Background] Chen CX, Kroenke K, Stump TE, Kean J, Carpenter JS, Krebs EE, Bair MJ, Damush TM, Monahan PO. Estimating minimally important differences for the PROMIS pain interference scales: results from 3 randomized clinical trials. Pain. 2018 Apr;159(4):775-782. doi: 10.1097/j.pain.0000000000001121. PMID 29200181
- [Background] Matheny AP, Wachs TD, Ludwig JL, Phillips K. Bringing order out of chaos: Psychometric characteristics of the confusion, hubbub, and order scale. J Appl Dev Psychol. 1995;16(3):429-444.
- [Background] Zullig LL, Shaw RJ, Crowley MJ, Lindquist J, Grambow SC, Peterson E, Shah BR, Bosworth HB. Association between perceived life chaos and medication adherence in a postmyocardial infarction population. Circ Cardiovasc Qual Outcomes. 2013 Nov;6(6):619-25. doi: 10.1161/CIRCOUTCOMES.113.000435. Epub 2013 Nov 12. PMID 24221839
- [Background] Jazowski SA, Sico IP, Lindquist JH, Smith VA, Bosworth HB, Danus S, Provenzale D, Kelley MJ, Zullig LL. Transportation as a barrier to colorectal cancer care. BMC Health Serv Res. 2021 Apr 13;21(1):332. doi: 10.1186/s12913-021-06339-x. PMID 33849524
- [Background] Drennan J. Cognitive interviewing: verbal data in the design and pretesting of questionnaires. J Adv Nurs. 2003 Apr;42(1):57-63. doi: 10.1046/j.1365-2648.2003.02579.x. PMID 12641812
- [Background] Willis GB. Cognitive interviewing: A tool for improving questionnaire design. Sage Publications; 2004.
- [Background] Willis GB, Artino AR Jr. What Do Our Respondents Think We're Asking? Using Cognitive Interviewing to Improve Medical Education Surveys. J Grad Med Educ. 2013 Sep;5(3):353-6. doi: 10.4300/JGME-D-13-00154.1. No abstract available. PMID 24404294
- [Background] Sandelowski M. Qualitative analysis: what it is and how to begin. Res Nurs Health. 1995 Aug;18(4):371-5. doi: 10.1002/nur.4770180411. PMID 7624531
- [Background] Guest, G., MacQueen, K.M. and Namey, E.E. (2012) Applied Thematic Analysis. Sage Publications, Inc., Thousand Oaks. http://www.sagepub.com/books/Book233379
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Background] Musselwhite K, Cuff L, McGregor L, King KM. The telephone interview is an effective method of data collection in clinical nursing research: a discussion paper. Int J Nurs Stud. 2007 Aug;44(6):1064-70. doi: 10.1016/j.ijnurstu.2006.05.014. Epub 2006 Jul 17. PMID 16844128
- [Background] Drabble L, Trocki KF, Salcedo B, Walker PC, Korcha RA. Conducting qualitative interviews by telephone: Lessons learned from a study of alcohol use among sexual minority and heterosexual women. Qual Soc Work. 2016 Jan;15(1):118-133. doi: 10.1177/1473325015585613. Epub 2016 May 14. PMID 26811696
- [Background] Creswell J, Plano Clark V. Designing & Conducting Mixed Methods Research. 2 ed. Thousand Oaks, CA: Sage; 2011.
- [Background] Lewinski AA, Anderson RA, Vorderstrasse AA, Fisher EB, Pan W, Johnson CM. Type 2 Diabetes Education and Support in a Virtual Environment: A Secondary Analysis of Synchronously Exchanged Social Interaction and Support. J Med Internet Res. 2018 Feb 21;20(2):e61. doi: 10.2196/jmir.9390. PMID 29467118
- [Result] Lewinski AA, Shapiro A, Crowley MJ, Whitfield C, Jones JR, Jeffreys AS, Coffman CJ, Howard T, McConnell E, Tanabe P, Barcinas S, Bosworth HB. Diabetes distress in Veterans with type 2 diabetes mellitus: Qualitative descriptive study. J Health Psychol. 2024 Dec;29(14):1593-1607. doi: 10.1177/13591053241233387. Epub 2024 Feb 21. PMID 38384142
- [Result] Lewinski AA, Shapiro A, Bosworth HB, Crowley MJ, McCant F, Howard T, Jeffreys AS, McConnell E, Tanabe P, Barcinas S, Coffman CJ, King HA. Veterans' Interpretation of Diabetes Distress in Diabetes Self-Management: Findings From Cognitive Interviews. Sci Diabetes Self Manag Care. 2021 Oct;47(5):391-403. doi: 10.1177/26350106211043487. Epub 2021 Sep 24. PMID 34559032

RESULTS

PARTICIPANT FLOW:
Groups:
- Aim 3b - TARDIS Intervention: Design & pilot test an innovative, tailored self-management information and supportive services intervention for Veterans with T2D, to promote engagement in self-management behaviors.
Period: Overall Study
Arm/Group | Aim 3a - TARDIS Photo Elicitation | Aim 3b - TARDIS Intervention
Started (Consented) | 14 | 20
Completed Baseline | 13 | 20
Completed | 3 | 18
Not Completed | 11 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 10 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aim 3a - TARDIS Photo Elicitation | Aim 3b - TARDIS Intervention | Total
Number analyzed (Participants) | 14 | 20 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.143 (10.918) | 64.4 (7.591) | 62.647 (9.201)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 9 | 17 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 7 | 16 | 23
  White | 4 | 4 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 12 | 19 | 31
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 20 | 34
Diabetes Distress Scale Score [Mean (Standard Deviation); unit: Total score] | 1.979 (0.781) | 1.824 (0.784) | 1.888 (0.775)

OUTCOME MEASURES:

1. Primary Outcome: Diabetes Distress Scale Score
Description: Scale used: 17 item Diabetes Distress Scale. Minimum value 1, Maximum value 6 Scoring is: < 2.0 is little or no distress; 2.0-2.9 is moderate distress; and ≥ 3.0 is high distress.
  Higher scores indicate higher diabetes distress or worse outcome.
Time Frame: Baseline
Population: For Aim 3a, participants did not complete a follow-up survey to assess their Diabetes Distress Scale score as this was not a part of the study design. Only participants in Aim3b (intervention) completed a baseline and follow-up survey to assess their DDS score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Aim 3a - TARDIS Photo Elicitation | Aim 3b - TARDIS Intervention
Number analyzed (Participants) | 14 | 20
score on a scale
  Baseline | 1.979 (0.781) | 1.824 (0.784)
  Follow-Up: number analyzed (Participants) | 0 | 20
  Follow-Up |  | 1.781 (0.653)

2. Primary Outcome: HbA1c Value
Description: The HbA1c value is determined from a blood test that measures a patient's average blood glucose level over the past 2 to 3 months.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin
Arm/Group | Aim 3a - TARDIS Photo Elicitation | Aim 3b - TARDIS Intervention
Number analyzed (Participants) | 14 | 20
percentage of glycosylated hemoglobin | 8.464 (2.367) | 9.705 (1.508)

3. Primary Outcome: Photo Elicitation (Aim 3a) Semi-Structured Interviews
Description: Number of semi-structured interviews completed by participants (1 interview per time point per participant)
Time Frame: From consent up to 1 month
Population: All participants who consent to Aim 3a will participate in this aim only. There is no randomization process or groups for this aim.
Measure: Number; unit: count of calls completed
Groups:
- Aim 3a - TARDIS Photo Elicitation: To further understand Diabetes Distress (DD) by expanding on what we have learned thus far in semi-structured interviews with Veterans. Visual-based qualitative methods will help identify and more robustly describe DD in Veterans.
Arm/Group | Aim 3a - TARDIS Photo Elicitation
Number analyzed (Participants) | 14
count of calls completed
  Consented | 14
  Baseline | 13
  Photo elicitation interview #1 | 5
  Photo elicitation interview #2 | 3

4. Secondary Outcome: Health Coaching Calls (Aim 3b - TARDIS Intervention)
Description: Number of Health Coaching Calls Completed (1 call per participant per time point)
Time Frame: Coaching calls started two weeks post-baseline to occur up to 3 months after consent
Population: All participants who consent to Aim 3b will participate in this aim only. There is no randomization process or groups for this aim.
Measure: Number; unit: Count of Calls Completed
Arm/Group | Aim 3b - TARDIS Intervention
Number analyzed (Participants) | 20
Count of Calls Completed
  Health Coaching Call #1 | 20
  Health Coaching Call #2 | 20
  Health Coaching Call #3 | 19

ADVERSE EVENTS:
Time Frame: From enrollment until study completion, up to 3 months
Arm/Group | Aim 3a - TARDIS Photo Elicitation | Aim 3b - TARDIS Intervention
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/20
Other Adverse Events (participants affected / at risk) | 0/14 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-30): https://cdn.clinicaltrials.gov/large-docs/51/NCT06972251/Prot_SAP_000.pdf